CLINICAL TRIAL: NCT01112020
Title: Components & Tolerability of Chlorhexidine Gluconate Dressing Patch Compared to BioPatch & Tegaderm Chlorhexidine Gluconate Securement Dressing After Application to Healthy Subjects Over a 7-day Period
Brief Title: Components of Chlorhexidine Gluconate Dressing
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: S10-0088
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: Chlorhexidine digluconate (CHG); Biopatch Protective Disk; Tegaderm CHG IV (intravenous) Securement Dressing; parachloroaniline (PCA); No condition being studied.; Assessing components of CHG-containing dressings after use.

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CHG Catheter Dressing Patch (Experimental)
  Interventions: Device: CHG Catheter Dressing Patch
- Biopatch (Active Comparator): Biopatch Protective Disk with CHG
  Interventions: Device: Biopatch
- Tegaderm CHG (Active Comparator): Tegaderm CHG IV Securement Dressing
  Interventions: Device: Tegaderm CHG

INTERVENTIONS:
Device: CHG Catheter Dressing Patch — 2% CHG dressing applied to 7 sites
  Arms: CHG Catheter Dressing Patch
Device: Biopatch — Biopatch applied to 7 sites
  Arms: Biopatch
Device: Tegaderm CHG — Tegaderm CHG IV Securement Dressing applied to 7 sites
  Arms: Tegaderm CHG

SUMMARY:
The purpose of this study is to determine the contents of a chlorhexidine-containing dressing after use.

DETAILED DESCRIPTION:
To characterize the chemical composition of the CHG (2% CHG) Catheter Dressing Patch as compared to Biopatch Protective Disk with CHG, and Tegaderm IV (intravenous) Securement Dressing over a wear period of 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Able to read, review and sign the Informed Consent
* Willing to shower using the same soap/cleansers from the Screening Visit through the end of the study
* Use study-approved contraceptive methods

Exclusion Criteria:

* Participation in an investigational study within 28 days prior to dosing.
* Clinically significant illness within 28 days prior to dosing.
* History of allergic responses to chlorhexidine, chlorhexidine-containing products, glycerol, adhesives, latex
* History of clinically significant skin disorders
* History of Type I diabetes mellitus, insulin-dependent diabetes mellitus(IDDM)
* History of significant dermatologic cancers (melanoma, squamous)
* Known history of immunologic disorders
* Use immunosuppressive or other proscribed medications
* Use of skin products at the application site
* Significant history of allergies to soaps, lotions, emollients, ointments, creams
* History of drug or alcohol addiction within the past year
* Pregnant, lactating, breast-feeding, or intends to become pregnant during the course of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Chlorhexidine gluconate (CHG) level | 1 week
  CHG level in dressing after 7 days exposure to CHG-containing test articles

SECONDARY OUTCOMES:
Parachloroaniline (PCA) level | 7 days
  PCA level in dressing after 7 days exposure to CHG-containing test articles

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Vargas, MD, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Saint Charles, Missouri, United States